CLINICAL TRIAL: NCT03499587
Title: Effects of Maternal Obesity on Offspring Brain Development
Status: Active, not recruiting | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 206551
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese pregnant women: BMI >30 with early OB visit medical records accessible
- Normal weight pregnant women: BMI 18.5-25 with early OB visit medical records accessible.

SUMMARY:
The goal of this study is to see if there are negative effects of maternal obesity during pregnancy on offspring's brain development.

DETAILED DESCRIPTION:
This study will recruit pregnant women who are either obese or normal weight and otherwise healthy. We will measure their body composition, food intake and other characteristics during pregnancy. When their babies are born, we will evaluate the brain development of their babies using magnetic resonance imaging and electroencephalography at age two weeks. We will then compare the findings and see if their are differences.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-25 or >30 with early OB visit medical records accessible
* singleton pregnancy
* about 36wks of pregnancy
* at least 18 years of age

Exclusion Criteria:

* hypertension, diabetes, or other preexisting medical conditions
* medications known to influence fetal growth
* recreational drugs, nicotine or tobacco use of alcohol use while pregnant
* pregnancy conception with assisted fertility treatment
* medical complications developed during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2026-06-27 (Estimated); Study Completion 2026-12-27 (Estimated)

PRIMARY OUTCOMES:
Determine whether maternal obesity correlates with abnormal brain development in newborns | 2 weeks
  Brain will be imaged at 2wks using an MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States